CLINICAL TRIAL: NCT07129707
Title: Does Nasal High-flow Oxygen Potentiate the Effects of Rehabilitative Exercise Training in Chronic Fibrotic Interstitial Lung Disease?
Brief Title: Nasal High-flow Oxygen Therapy During Acute Exercise in Fibrotic Interstitial Lung Disease
Acronym: PID-OXacute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dieulefit Santé Centre de Réadaptation (Other)
Responsible Party: Principal Investigator, Frédéric Hérengt, Principal Investigator, Dieulefit Santé Centre de Réadaptation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: DieulefitSante
Record Dates: First submitted 2025-08-09; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Lung Disease (ILD)
Keywords: Dyspnea; Exercise; Oxygen inhalation therapy; Pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Dyspnea; Motor Activity; Pulmonary Fibrosis | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Crossover - 4 experimental conditions
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Room Air (Placebo Comparator): Room Air breathing (flow= 0 L/min; inspired fraction of O2= 0.21)
  Interventions: Other: Exercise testing
- Supplemental Oxygen (Active Comparator): Supplemental oxygen therapy (flow= 9-12 L/min; inspired fraction of O2= 1.0)
  Interventions: Other: Exercise testing
- Nasal high-flow (Active Comparator): Nasal high-flow (flow= 50-70 L/min; inspired fraction of O2= 0.21)
  Interventions: Other: Exercise testing
- Nasal high-flow oxygen therapy (Active Comparator): Nasal high-flow oxygen therapy (flow= 50-70 L/min; inspired fraction of O2= 0.50)
  Interventions: Other: Exercise testing

INTERVENTIONS:
Other: Exercise testing — Each participant performs a constant work-rate exercise test (70% peak work rate) under the 4 experimental conditions (referred as arms).

SUMMARY:
Hallmarks of fibrotic interstitial lung disease (f-ILD) include severe hypoxemia, dyspnea and exercise limitation. Although ambulatory oxygen (O2) therapy is widely prescribed, standard low-flow O2 systems (nasal prongs) fail to meet patients' inspiratory demand on exertion resulting in incomplete correction of hypoxemia and limited symptomatic relief. Nasal high-flow O2 therapy (NHFO2) delivers heated, humidified, and O2-enriched air at high flow rates. It has recently emerged as a promising alternative to overcome the pre-specified limitations: NHFO2 is more effective in correcting hypoxemia and reducing dyspnea vs standard O2 therapy and consistently improved exercise capacity in f-ILD. In fact, NHF per se may exert independent physiological benefits such as washout of the anatomical dead space and reduced work of breathing. However, the respective effect of respiratory support and improved oxygenation on dyspnea and exercise tolerance remain unexplored in f-ILD. To address this gap in knowledge, this prospective, randomized-controlled trial aimed to disentangle the i) independent and ii) combined effects of respiratory support and supplemental O2 on dyspnea and exercise tolerance in patients with f-ILD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibrotic interstitial lung disease (regardless of etiology)
* age ≥18 years
* modified Medical Research Council scale ≥1
* stable condition (no acute exacerbation within the preceding 3 months)

Exclusion Criteria:

* inability to perform a cardiopulmonary exercise test (CPET) on a bicycle ergometer
* participation in a pulmonary rehabilitation program within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Time to exercise intolerance | 4 times over 2 consecutive days (1 time per experimental condition)
  Measured during a constant work-rate exercise test (70% peak work rate)
Isotime dyspnea | 4 times over 2 consecutive days (1 time per experimental condition)
  0-10 category-ratio Borg scale

SECONDARY OUTCOMES:
Breathing pattern | 4 times over 2 consecutive days (1 time per experimental condition)
  Respiratory inductive plethysmography
Gas exchange | 4 times over 2 consecutive days (1 time per experimental condition)
  Earlobe capnography
Quadriceps muscle oxygenation | 4 times over 2 consecutive days (1 time per experimental condition)
  Near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Marillier, PhD, Study Chair — University Grenoble Alps
Locations (1):
- Centre de Réadaptation Cardio-Respiratoire Dieulefit Santé, Dieulefit, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be available from the contact person on reasonable request.

REFERENCES:
- [Background] Girault C, Boyer D, Jolly G, Carpentier D, Beduneau G, Frat JP. [Operating principles, physiological effects and practical issues of high-flow nasal oxygen therapy]. Rev Mal Respir. 2022 May;39(5):455-468. doi: 10.1016/j.rmr.2022.03.012. Epub 2022 May 16. French. PMID 35589480
- [Background] Badenes-Bonet D, Cejudo P, Rodo-Pin A, Martin-Ontiyuelo C, Chalela R, Rodriguez-Portal JA, Vazquez-Sanchez R, Gea J, Duran X, Caguana OA, Rodriguez-Chiaradia DA, Balcells E. Impact of high-flow oxygen therapy during exercise in idiopathic pulmonary fibrosis: a pilot crossover clinical trial. BMC Pulm Med. 2021 Nov 8;21(1):355. doi: 10.1186/s12890-021-01727-9. PMID 34749699
- [Background] Harada J, Nagata K, Morimoto T, Iwata K, Matsunashi A, Sato Y, Tachikawa R, Ishikawa A, Tomii K. Effect of high-flow nasal cannula oxygen therapy on exercise tolerance in patients with idiopathic pulmonary fibrosis: A randomized crossover trial. Respirology. 2022 Feb;27(2):144-151. doi: 10.1111/resp.14176. Epub 2021 Nov 2. PMID 34729862
- [Background] Al Chikhanie Y, Veale D, Verges S, Herengt F. The effect of heated humidified nasal high flow oxygen supply on exercise tolerance in patients with interstitial lung disease: A pilot study. Respir Med. 2021 Sep;186:106523. doi: 10.1016/j.rmed.2021.106523. Epub 2021 Jun 29. PMID 34225230
- [Background] Jacobs SS, Krishnan JA, Lederer DJ, Ghazipura M, Hossain T, Tan AM, Carlin B, Drummond MB, Ekstrom M, Garvey C, Graney BA, Jackson B, Kallstrom T, Knight SL, Lindell K, Prieto-Centurion V, Renzoni EA, Ryerson CJ, Schneidman A, Swigris J, Upson D, Holland AE. Home Oxygen Therapy for Adults with Chronic Lung Disease. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2020 Nov 15;202(10):e121-e141. doi: 10.1164/rccm.202009-3608ST. PMID 33185464